CLINICAL TRIAL: NCT05568797
Title: A Phase III, Open-label, Randomized, Controlled, Multi-country Study to Evaluate the Immune Response, Safety and Reactogenicity of an RSVPreF3 OA Investigational Vaccine When Co-administered With FLU aQIV (Inactivated Influenza Vaccine - Adjuvanted) in Adults Aged 65 Years and Above
Brief Title: A Study on the Immune Response and Safety of a Vaccine Against Respiratory Syncytial Virus (RSV) When Given Alone or Co-administered With an Adjuvanted Vaccine Against Influenza in Adults Aged 65 Years and Above
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 218350; 2022-000623-21 (EudraCT Number)
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory syncytial virus; Adjuvanted quadrivalent influenza vaccine; Immunogenicity; Safety; Reactogenicity; Adults aged 65 years and above
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Co-Ad Group (Experimental): Participants received one dose of FLU-aQIV vaccine and one dose of RSVPreF3 OA vaccine, both doses administered at Day 1, and were followed until end of study.
  Interventions: Biological: RSVPreF3 OA vaccine; Biological: FLU vaccine
- Control Group (Active Comparator): Participants received one dose of FLU-aQIV vaccine at Day 1, followed by one dose of RSVPreF3 OA vaccine at Day 31, and were followed until end of study.
  Interventions: Biological: RSVPreF3 OA vaccine; Biological: FLU vaccine

INTERVENTIONS:
Biological: RSVPreF3 OA vaccine — One dose of RSVPreF3 OA vaccine administered intramuscularly.
Biological: FLU vaccine — One dose of FLU vaccine administered intramuscularly.
  Other Names: Fluad Tetra, FLUAD QUADRIVALENT, Fluad Quad

SUMMARY:
The aim of this study is to assess the immunogenicity, safety and reactogenicity of the RSV PreFusion protein 3 older adult (RSVPreF3 OA) investigational vaccine when co-administered with an adjuvanted quadrivalent influenza (FLU aQIV) vaccine, in adults aged 65 years of age (YOA).

ELIGIBILITY:
Inclusion Criteria:

* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of the electronic diary cards [eDiaries], return for follow-up visits, ability to access and utilize a phone or other electronic communications).
* A male or female ≥ 65 YOA at the time of the first study intervention administration.
* Participants living in the general community or in an assisted-living facility that provides minimal assistance, such that the participant is primarily responsible for self-care and activities of daily living.
* Written or witnessed informed consent obtained from the participant prior to performance of any study-specific procedure.
* Participants who are medically stable in the opinion of the investigator at the time of first study intervention administration. Participants with chronic stable medical conditions with or without specific treatment, such as diabetes, hypertension or cardiac disease, are allowed to participate in this study if considered by the investigator as medically stable.

Exclusion Criteria:

Medical conditions

* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease or immunosuppressive/cytotoxic therapy, based on medical history and physical examination (no laboratory testing required).
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study interventions, in particular any history of severe allergic reaction to egg protein or to a previous influenza vaccine.
* Hypersensitivity to latex.
* Guillain-Barré syndrome that occurred within 6 weeks of receipt of prior influenza vaccine.
* Serious or unstable chronic illness.
* Any history of dementia or any medical condition that moderately or severely impairs cognition.
* Recurrent or uncontrolled neurological disorders or seizures. Participants with medically-controlled active or chronic neurological diseases can be enrolled in the study as per investigator assessment, provided that their condition will allow them to comply with the requirements of the protocol.
* Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.

Prior/Concomitant therapy

* Use of any investigational or non-registered product (drug, vaccine, or medical device) other than the study interventions during the period beginning 30 days before the first dose of study interventions, or planned use during the study period.
* Administration of an influenza vaccine during the 6 months preceding the study FLU vaccine administration.
* Planned or actual administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first study intervention administration and ending 30 days after the last study intervention administration. In the case of COVID-19 vaccines, this time window can be decreased to 14 days before and after each study intervention administration provided this COVID-19 vaccine use is in line with local governmental recommendations.
* Previous vaccination with an RSV vaccine.
* Administration of long-acting immune-modifying drugs or planned administration at any time during the study period.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 90 days before the administration of first dose of study interventions or planned administration during the study period.
* Chronic administration (defined as more than 14 consecutive days in total) of immunosuppressants or other immune-modifying drugs during the period starting 90 days prior to the first study intervention dose or planned administration during the study period. For corticosteroids, this will mean prednisone ≥ 20 mg/day, or equivalent. Inhaled and topical steroids are allowed.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product (drug or invasive medical device).

Other exclusions

* History of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential participant unable/unlikely to provide accurate safety reports or comply with study procedures.
* Bedridden participants.
* Planned move during the study conduct that prohibits participation until study end.
* Participation of any study personnel or their immediate dependents, family, or household members.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1045 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-07-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- Belgium (4):
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Erpent
  - GSK Investigational Site, Genk
  - GSK Investigational Site, Ieper
- Finland (6):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
- France (8):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nîmes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pierre-Bénite
- Spain (11):
  - GSK Investigational Site, Marbella - Málaga, Andalusia
  - GSK Investigational Site, Benalmádena, Málaga
  - GSK Investigational Site, Boadilla Del Monte (Madrid)
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Centelles
  - GSK Investigational Site, La Roca Del Valles (Barcelona)
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Salamanca
  - GSK Investigational Site, Santander (Cantabria)
  - GSK Investigational Site, Valladolid
  - GSK Investigational Site, Vic
- United Kingdom (7):
  - GSK Investigational Site, Soham, Cambridgeshire
  - GSK Investigational Site, Bollington, Cheshire
  - GSK Investigational Site, Chippenham, Wiltshire
  - GSK Investigational Site, Blackpool
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Chippenham
  - GSK Investigational Site, Peterborough

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data (IPD) and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Background] Clark R, Davies S, Labrador J, Loubet P, Natalini Martinez S, Morinigo HM, Nicolas JF, Vera MP, Ramet M, Rebollo-Rodrigo MH, Sanz-Munoz I, Dezutter N, Germain S, David MP, Jayadev A, Amare Hailemariam H, Kotb S, Meyer N. Safety and Immunogenicity of Respiratory Syncytial Virus Prefusion F Protein Vaccine when Co-administered with Adjuvanted Seasonal Quadrivalent Influenza Vaccine in Older Adults: A Phase 3 Randomized Trial. Clin Infect Dis. 2024 Oct 15;79(4):1088-1098. doi: 10.1093/cid/ciae365. PMID 39099085

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All 1045 enrolled participants were randomized to Co-Ad and Control Groups and received at least 1 dose of study intervention and were included in the exposed set.
Pre-assignment Details: This study assessed the immunogenicity, safety and reactogenicity of the RSVPre3 OA vaccine when co-administered with an adjuvanted quadrivalent influenza (FLU-aQIV [FLU]) vaccine, in adults aged 65 years old or above.
Period: Overall Study
Arm/Group | Co-Ad Group | Control Group
Started | 523 | 522
Completed | 518 | 499
Not Completed | 5 | 23
Not completed — Adverse Event | 0 | 8
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 1 | 10
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Co-Ad Group | Control Group | Total
Number analyzed (Participants) | 523 | 522 | 1045
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 72.1 (5.4) | 72.2 (5.2) | 72.2 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 255 | 275 | 530
  Male | 268 | 247 | 515
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 0 | 1 | 1
  Black or African American | 0 | 1 | 1
  White | 522 | 516 | 1038
  Multiple | 0 | 1 | 1
  Other - Unspecified | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Titers for Hemagglutination Inhibition (HI) Antibodies Against 4 FLU Vaccine Strains Expressed as Group Geometric Mean Titers (GMTs) at 1 Month After FLU Vaccine Dose
Description: HI antibodies assessed were antibodies against the Flu A/Darwin/6/2021 H3N2, Flu A/Victoria/2570/2019 H1N1, Flu B/Austria/1359417/2021 Victoria, and Flu B/Phuket/3073/2013 Yamagata flu strains.
Time Frame: At 1 month after the FLU vaccine dose (Day 31 for both groups)
Population: Analysis was performed on Per Protocol Set for FLU analysis which included eligible participants who: received at least one control group intervention or all Co-Ad group interventions, had pre- and post-dose immunogenicity results, adhered to specified blood draw intervals, with immunogenicity data available for the specified analysis at the specified time point post-FLU vaccine dose, who lacked interfering medical conditions and avoided prohibited concomitant medication/vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 429 | 400
Titers
  Flu A/Darwin/6/2021 H3N2 | 43.8 [38.9 to 49.4] | 57.7 [51.0 to 65.3]
  Flu A/Victoria/2570/2019 H1N1: number analyzed (Participants) | 420 | 396
  Flu A/Victoria/2570/2019 H1N1 | 143.0 [128.6 to 159.0] | 148.5 [133.2 to 165.6]
  Flu B/Austria/1359417/2021 Victoria | 613.9 [575.1 to 655.2] | 597.5 [558.7 to 639.1]
  Flu B/Phuket/3073/2013 Yamagata: number analyzed (Participants) | 428 | 400
  Flu B/Phuket/3073/2013 Yamagata | 406.2 [380.0 to 434.2] | 421.0 [393.0 to 451.0]
Statistical Analysis 1: Comparison: Co-Ad Group vs Control Group; To demonstrate the non-inferiority of the FLU vaccine when co administered with the RSVPreF3 OA vaccine compared to the FLU vaccine administered alone, in terms of HI GMTs against the Flu A/Darwin/6/2021 H3N2 strain, at 1 month post-FLU vaccine dose administration (Day 31 for both groups); Test type: Non-Inferiority — The non-inferiority is demonstrated if the upper limit (UL) of the 2-sided 95% confidence interval (CI) of the group GMT ratio (Control group divided by Co-Ad group) for HI antibody titers for the Flu strain is less than or equal (<=) 1.5; GMT Ratio = 1.32, 0.95% CI 2-sided [1.13 to 1.53] — The comparison was done using adjusted group ratio of GMT (ANCOVA model applied to the logarithm- transformed titers). The ANCOVA model included the treatment group and the age category as fixed effects and the pre-dose log-10 titer as covariate
Statistical Analysis 2: Comparison: Co-Ad Group vs Control Group; To demonstrate the non-inferiority of the FLU vaccine when co administered with the RSVPreF3 OA vaccine compared to the FLU vaccine administered alone, in terms of HI GMTs against the Flu A/Victoria/2570/2019 H1N1 influenza strain included in the FLU vaccine, at 1 month post-FLU vaccine dose administration (Day 31 for both groups); Test type: Non-Inferiority — The non-inferiority is demonstrated if the UL of the 2-sided 95% CI of the group GMT ratio (Control group divided by Co-Ad group) for HI antibody titers for the Flu strain is <=1.5; GMT Ratio = 1.04, 0.95% CI 2-sided [0.91 to 1.18] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Co-Ad Group vs Control Group; To demonstrate the non-inferiority of the FLU vaccine when co administered with the RSVPreF3 OA vaccine compared to the FLU vaccine administered alone, in terms of HI GMTs against the Flu B/Austria/1359417/2021 influenza strain included in the FLU vaccine, at 1 month post-FLU vaccine dose administration (Day 31 for both groups); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT Ratio = 0.97, 0.95% CI 2-sided [0.90 to 1.06] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Co-Ad Group vs Control Group; To demonstrate the non-inferiority of the FLU vaccine when co administered with the RSVPreF3 OA vaccine compared to the Flu vaccine administered alone, in terms of HI GMTs against the Flu B/Phuket/3073/2013 Yamagata influenza strain included in the FLU vaccine, at 1 month post-FLU vaccine dose administration (Day 31 for both groups); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT Ratio = 1.04, 0.95% CI 2-sided [0.95 to 1.13] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: RSV-A Neutralizing Antibody Titers Expressed as GMTs
Description: RSV-A neutralizing antibodies were given as GMTs and expressed as Estimated Dilution 60 (ED60).
Time Frame: At 1 month after the RSVPreF3 OA dose (Day 31 for the Co-Ad Group and Day 61 for the Control Group)
Population: Analysis was performed on Per Protocol Set for RSV OA analysis which included eligible participants who: received at least one control group intervention or all Co-Ad group interventions, had pre- and post-dose immunogenicity results, adhered to specified blood draw intervals, with immunogenicity data available for the specified analysis at the specified time point post-RSVPreF3 OA vaccine dose, who lacked interfering medical conditions and avoided prohibited concomitant medication/vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 471 | 373
Titers | 6673.4 [6057.2 to 7352.4] | 6591.8 [5917.8 to 7342.6]
Statistical Analysis 1: Comparison: Co-Ad Group vs Control Group; To demonstrate the non-inferiority of the RSVPreF3 OA vaccine when co-administered with the FLU vaccine compared to the RSVPreF3 OA vaccine administered alone, in terms of RSV-A neutralizing antibody titers, at 1 month after the RSVPreF3 OA vaccine dose (Day 31 for the Co-Ad Group and Day 61 for the Control Group); Test type: Non-Inferiority — The non-inferiority is demonstrated if the UL of the 2-sided 95% CI of the GMT ratio (Control group divided by Co-Ad group) for RSV-A neutralizing antibody vaccine is <=1.5; GMT Ratio = 0.99, 0.95% CI 2-sided [0.87 to 1.12] — The comparison is done using adjusted group ratio of GMT (ANCOVA model applied to the logarithm- transformed titers). The ANCOVA model included the treatment group and the age category as fixed effects and the pre-dose log-10 titer as covariate

3. Primary Outcome: RSV-B Neutralizing Antibody Titers Expressed as GMTs
Description: RSV B neutralizing antibodies are given as GMTs and expressed as Estimated Dilution 60 (ED60).
Time Frame: At 1 month after the RSVPreF3 OA dose (Day 31 for the CoAd Group and Day 61 for the Control Group)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 469 | 373
Titers | 7880.1 [7195.4 to 8629.8] | 9134.1 [8255.9 to 10105.7]
Statistical Analysis 1: Comparison: Co-Ad Group vs Control Group; To demonstrate the non-inferiority of the RSVPreF3 OA vaccine when co-administered with the FLU vaccine compared to the RSVPreF3 OA vaccine administered alone, in terms of RSV-B neutralizing antibody titers, at 1 month after the RSVPreF3 OA vaccine dose (Day 31 for the CoAd Group and Day 61 for the Control Group); Test type: Non-Inferiority — The non-inferiority is demonstrated if the UL of the 2-sided 95% CI of the GMT ratio (Control group divided by Co-Ad group) for RSV-B neutralizing antibody vaccine is <=1.5; GMT Ratio = 1.16, 0.95% CI 2-sided [1.03 to 1.30] — The comparison is done using adjusted group ratio of GMT (ANCOVA model applied to the logarithm- transformed titers). The ANCOVA model included the treatment group, the age category as fixed effects and the pre-dose log-10 titer as covariate

4. Secondary Outcome: HI Seroconversion Rate (SCR) for 4 FLU Vaccine Strains
Description: SCR for HI antibody is defined as the percentage of participants who have either a HI predose titer less than (<) 1:10 and a post-dose titer greater than or equal to (>=) 1:40, or a pre-dose titer >= 1:10 and at least a 4-fold increase in post-dose titer. The assessed Flu strains were: Flu A/Darwin/6/2021 H3N2, Flu A/Victoria/2570/2019 H1N1, Flu B/Austria/1359417/2021 Victoria, and Flu B/Phuket/3073/2013 Yamagata.
Time Frame: At 1 month after the FLU vaccine dose (Day 31 for both groups)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 429 | 400
Percentage of participants
  Flu A/Darwin/6/2021 H3N2 | 51.7 [46.9 to 56.6] | 62.0 [57.0 to 66.8]
  Flu A/Victoria/2570/2019 H1N1: number analyzed (Participants) | 420 | 396
  Flu A/Victoria/2570/2019 H1N1 | 44.0 [39.2 to 48.9] | 45.7 [40.7 to 50.8]
  Flu B/Austria/1359417/2021 Victoria | 17.2 [13.8 to 21.2] | 17.5 [13.9 to 21.6]
  Flu B/Phuket/3073/2013 Yamagata: number analyzed (Participants) | 428 | 400
  Flu B/Phuket/3073/2013 Yamagata | 18.5 [14.9 to 22.5] | 19.3 [15.5 to 23.5]
Statistical Analysis 1: Comparison: Co-Ad Group vs Control Group; To evaluate the non-inferiority of the FLU vaccine when co-administered with the RSVPreF3 OA vaccine compared to the FLU vaccine administered alone as measured by the difference of percentage of participants achieving seroconversion for HI antibody titers against Flu A/Darwin/6/2021 H3N2 strain at 1 month post-FLU vaccine dose administration (Day 31 for both groups); Test type: Non-Inferiority — The non-inferiority is demonstrated if the UL of the 2-sided 95% CI on the group difference (Control group minus Co-Ad group) in terms of SCR is <=10% for anti-HI antibodies; Difference of Percentage = 10.25, 0.95% CI 2-sided [3.50 to 16.90]
Statistical Analysis 2: Comparison: Co-Ad Group vs Control Group; To evaluate the non-inferiority of the FLU vaccine when co-administered with the RSVPreF3 OA vaccine compared to the FLU vaccine administered alone as measured by the difference of percentage of participants achieving seroconversion for HI antibody titers against Flu A/Victoria/2570/2019 H1N1 strain at 1 month post-FLU vaccine dose administration (Day 31 for both groups); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Difference of Percentage = 1.66, 0.95% CI 2-sided [-5.16 to 8.47]
Statistical Analysis 3: Comparison: Co-Ad Group vs Control Group; To evaluate the non-inferiority of the FLU vaccine when co-administered with the RSVPreF3 OA vaccine compared to the FLU vaccine administered alone as measured by the difference of percentage of participants achieving seroconversion for HI antibody titers against Flu B/Austria/1359417/2021 Victoria at 1 month post-FLU vaccine dose administration (Day 31 for both groups); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Difference of Percentage = 0.25, 0.95% CI 2-sided [-4.92 to 5.46]
Statistical Analysis 4: Comparison: Co-Ad Group vs Control Group; To evaluate the non-inferiority of the FLU vaccine when co-administered with the RSVPreF3 OA vaccine compared to the FLU vaccine administered alone as measured by the difference of percentage of participants achieving seroconversion for HI antibody titers against Flu B/Phuket/3073/2013 Yamagata strain at 1 month post-FLU vaccine dose administration (Day 31 for both groups); Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Difference of Percentage = 0.79, 0.95% CI 2-sided [-4.54 to 6.17]

5. Secondary Outcome: RSV-A Neutralization Antibody Titers Expressed as Mean Geometric Increase (MGI)
Description: MGI was defined as the geometric mean of the within-participant ratios of the post-dose titer over the pre-dose titer.
Time Frame: At 1 month after the RSVPreF3 OA vaccine dose (Day 31 for the Co-Ad Group and Day 61 for the Control Group) compared to pre-vaccination (Day 1 for Co-Ad group and Day 31 for Control group)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 471 | 373
Ratio | 8.50 [7.79 to 9.27] | 7.58 [6.82 to 8.42]

6. Secondary Outcome: RSV-B Neutralization Antibody Titers Expressed as MGI
Description: MGI was defined as the geometric mean of the within-participant ratios of the post-dose titer over the pre-dose titer.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 469 | 373
Ratio | 7.11 [6.55 to 7.72] | 7.46 [6.74 to 8.25]

7. Secondary Outcome: Titers for HI Antibodies Against 4 FLU Vaccine Strains
Description: HI antibodies assessed were antibodies against the Flu A/Darwin/6/2021 H3N2, Flu A/Victoria/2570/2019 H1N1, Flu B/Austria/1359417/2021 Victoria, and Flu B/Phuket/3073/2013 Yamagata flu strains. HI antibodies were expressed as GMT, in titers.
Time Frame: At Day 1 (Baseline) and Day 31
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 469 | 449
Titers
  Flu A/Darwin/6/2021 H3N2, Day 1 | 9.1 [8.4 to 9.8] | 8.7 [8.1 to 9.4]
  Flu A/Darwin/6/2021 H3N2 , Day 31: number analyzed (Participants) | 442 | 400
  Flu A/Darwin/6/2021 H3N2 , Day 31 | 45.3 [40.6 to 50.5] | 58.3 [51.6 to 65.8]
  Flu A/Victoria/2570/2019 H1N1, Day 1: number analyzed (Participants) | 460 | 446
  Flu A/Victoria/2570/2019 H1N1, Day 1 | 40.0 [35.4 to 45.1] | 43.2 [38.4 to 48.5]
  Flu A/Victoria/2570/2019 H1N1, Day 31: number analyzed (Participants) | 440 | 399
  Flu A/Victoria/2570/2019 H1N1, Day 31 | 151.0 [136.4 to 167.2] | 163.8 [147.5 to 181.9]
  Flu B/Austria/1359417/2021 Victoria, Day 1 | 323.6 [300.4 to 348.5] | 327.2 [303.6 to 352.7]
  Flu B/Austria/1359417/2021 Victoria, Day 31: number analyzed (Participants) | 442 | 400
  Flu B/Austria/1359417/2021 Victoria, Day 31 | 614.9 [575.5 to 657.0] | 608.1 [566.8 to 652.5]
  Flu B/Phuket/3073/2013 Yamagata, Day 1: number analyzed (Participants) | 468 | 449
  Flu B/Phuket/3073/2013 Yamagata, Day 1 | 213.1 [198.5 to 228.7] | 193.2 [179.9 to 207.5]
  Flu B/Phuket/3073/2013 Yamagata, Day 31: number analyzed (Participants) | 442 | 400
  Flu B/Phuket/3073/2013 Yamagata, Day 31 | 423.0 [394.6 to 453.5] | 417.5 [387.9 to 449.4]

8. Secondary Outcome: HI Seroprotection Rate (SPR) for 4 FLU Vaccine Strains
Description: SPR for HI antibody was defined as the percentage of participants with a serum HI titer >= 1:40. The assessed Flu strains were: Flu A/Darwin/6/2021 H3N2, Flu A/Victoria/2570/2019 H1N1, Flu B/Austria/1359417/2021 Victoria, and Flu B/Phuket/3073/2013 Yamagata.
Time Frame: At Day 1 (Baseline) and Day 31
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 469 | 449
Percentage of participants
  Flu A/Darwin/6/2021 H3N2, Day 1 | 10.4 [7.8 to 13.6] | 10.7 [8.0 to 13.9]
  Flu A/Darwin/6/2021 H3N2, Day 31: number analyzed (Participants) | 442 | 400
  Flu A/Darwin/6/2021 H3N2, Day 31 | 63.6 [58.9 to 68.1] | 71.0 [66.3 to 75.4]
  Flu A/Victoria/2570/2019 H1N1, Day 1: number analyzed (Participants) | 460 | 446
  Flu A/Victoria/2570/2019 H1N1, Day 1 | 60.0 [55.4 to 64.5] | 64.3 [59.7 to 68.8]
  Flu A/Victoria/2570/2019 H1N1, Day 31: number analyzed (Participants) | 440 | 399
  Flu A/Victoria/2570/2019 H1N1, Day 31 | 92.0 [89.1 to 94.4] | 95.2 [92.7 to 97.1]
  Flu B/Austria/1359417/2021 Victoria, Day 1 | 99.6 [98.5 to 99.9] | 100 [99.2 to 100]
  Flu B/Austria/1359417/2021 Victoria, Day 31: number analyzed (Participants) | 442 | 400
  Flu B/Austria/1359417/2021 Victoria, Day 31 | 100 [99.2 to 100] | 100 [99.1 to 100]
  Flu B/Phuket/3073/2013 Yamagata, Day 1: number analyzed (Participants) | 468 | 449
  Flu B/Phuket/3073/2013 Yamagata, Day 1 | 99.8 [98.8 to 100.0] | 98.9 [97.4 to 99.6]
  Flu B/Phuket/3073/2013 Yamagata, Day 31: number analyzed (Participants) | 442 | 400
  Flu B/Phuket/3073/2013 Yamagata, Day 31 | 100 [99.2 to 100] | 100 [99.1 to 100]

9. Secondary Outcome: HI Antibody Titers for 4 FLU Vaccine Strains Expressed as MGI
Description: MGI was defined as the geometric mean of the within-participant ratios of the post-dose titer over the pre-dose titer. The assessed Flu strains were: Flu A/Darwin/6/2021 H3N2, Flu A/Victoria/2570/2019 H1N1, Flu B/Austria/1359417/2021 Victoria, and Flu B/Phuket/3073/2013 Yamagata.
Time Frame: At 1 month after the FLU dose (Day 31 for both groups) compared to pre-vaccination (Day 1 for both groups)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 429 | 400
Ratio
  Flu A/Darwin/6/2021 H3N2 HI | 5.10 [4.60 to 5.66] | 6.87 [6.12 to 7.71]
  Flu A/Victoria/2570/2019 H1N1 HI: number analyzed (Participants) | 420 | 396
  Flu A/Victoria/2570/2019 H1N1 HI | 3.85 [3.40 to 4.35] | 3.79 [3.34 to 4.31]
  Flu B/Austria/1359417/2021 Victoria HI | 1.89 [1.77 to 2.03] | 1.84 [1.71 to 1.98]
  Flu B/Phuket/3073/2013 Yamagata HI: number analyzed (Participants) | 428 | 400
  Flu B/Phuket/3073/2013 Yamagata HI | 1.94 [1.82 to 2.07] | 2.11 [1.97 to 2.27]

10. Secondary Outcome: Percentage of Participants Reporting Each Solicited Administration Site Event After Each Vaccine Dose Administration
Description: The solicited administration site events after vaccination include erythema, pain and swelling.
Time Frame: Within 7 days (the day of vaccination and 6 subsequent days) after each vaccine administration (vaccines administered at Day 1 for CoAd Group and at Day 1 and Day 31 for Control group)
Population: Analysis was performed on Exposed set which included participants who received a study intervention and with the electronic diary completed post-each vaccination and for whom solicited administration event data was available for specific visit. The Control group received FLU vaccination at Day 1 and RSVPreF3 OA vaccination at Day 31; Co-Ad group received co-administered vaccine (RSVPreF3 OA + FLU) on Day 1. Analysis per group is based on the study intervention administered on specific visit.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 516 | 513
Percentage of participants
  Erythema, FLU dose given at Day 1 | 6.6 [4.6 to 9.1] | 5.3 [3.5 to 7.6]
  Erythema, RSV dose given at Day 1: number analyzed (Participants) | 516 | 0
  Erythema, RSV dose given at Day 1 | 14.1 [11.3 to 17.5] |
  Erythema, RSV dose given at Day 31: number analyzed (Participants) | 0 | 451
  Erythema, RSV dose given at Day 31 |  | 12.4 [9.5 to 15.8]
  Pain, FLU dose given at Day 1 | 51.7 [47.3 to 56.1] | 44.8 [40.5 to 49.3]
  Pain, RSV dose given at Day 1: number analyzed (Participants) | 516 | 0
  Pain, RSV dose given at Day 1 | 66.1 [61.8 to 70.2] |
  Pain, RSV dose given at Day 31: number analyzed (Participants) | 0 | 451
  Pain, RSV dose given at Day 31 |  | 58.8 [54.1 to 63.3]
  Swelling, FLU dose given at Day 1 | 5.2 [3.5 to 7.5] | 6.0 [4.1 to 8.5]
  Swelling, RSV dose given at Day 1: number analyzed (Participants) | 516 | 0
  Swelling, RSV dose given at Day 1 | 10.5 [8.0 to 13.4] |
  Swelling, RSV dose given at Day 31: number analyzed (Participants) | 0 | 451
  Swelling, RSV dose given at Day 31 |  | 8.4 [6.0 to 11.4]

11. Secondary Outcome: Percentage of Participants Reporting Each Solicited Systemic Event After Each Dose Administration
Description: The solicited systemic events after vaccination include fever, headache, fatigue, myalgia and arthralgia.
Time Frame: Within 7 days (the day of vaccination and 6 subsequent days) after each vaccine administration (vaccines administered at Day 1 and Day 31 for C-oAd Group and at Day 1 and Day 31 for Control group)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 516 | 513
Percentage of participants
  Arthralgia, Dosing at Day 1 | 25.8 [22.1 to 29.8] | 15.6 [12.6 to 19.0]
  Arthralgia, Dosing at Day 31: number analyzed (Participants) | 0 | 451
  Arthralgia, Dosing at Day 31 |  | 17.1 [13.7 to 20.9]
  Fatigue, Dosing at Day 1 | 45.7 [41.4 to 50.1] | 28.5 [24.6 to 32.6]
  Fatigue, Dosing at Day 31: number analyzed (Participants) | 0 | 451
  Fatigue, Dosing at Day 31 |  | 30.4 [26.2 to 34.9]
  Fever, Dosing at Day 1 | 2.1 [1.1 to 3.8] | 0.6 [0.1 to 1.7]
  Fever, Dosing at Day 31: number analyzed (Participants) | 0 | 451
  Fever, Dosing at Day 31 |  | 1.1 [0.4 to 2.6]
  Headache, Dosing at Day 1 | 32.2 [28.2 to 36.4] | 19.3 [16.0 to 23.0]
  Headache, Dosing at Day 31: number analyzed (Participants) | 0 | 451
  Headache, Dosing at Day 31 |  | 23.9 [20.1 to 28.2]
  Myalgia, Dosing at Day 1 | 39.0 [34.7 to 43.3] | 23.0 [19.4 to 26.9]
  Myalgia, Dosing at Day 31: number analyzed (Participants) | 0 | 451
  Myalgia, Dosing at Day 31 |  | 31.9 [27.6 to 36.5]

12. Secondary Outcome: Percentage of Participants Reporting Unsolicited Adverse Events (AEs)
Description: An unsolicited AEs is an AE that is not included in a list of solicited events using a Participant Electronic Diary. Unsolicited events must be spontaneously communicated by a participant who signs the informed consent. Unsolicited AEs include both serious, non-serious AEs and potential immune-mediated diseases (pIMDs).
Time Frame: Within 30 days (the day of vaccination and 29 subsequent days) after each vaccine administration
Population: Analysis was performed on Exposed set which included participants who received at least a study intervention and had data for the assessed timepoint and analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 523 | 522
Percentage of participants | 13.6 [10.8 to 16.8] | 24.5 [20.9 to 28.4]

13. Secondary Outcome: Percentage of Participants Reporting at Least One Serious Adverse Event (SAEs)
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, or results in disability/incapacity or is a congenital anomaly/birth defect in the offspring of a study participant.
Time Frame: From Day 1 until 6 months after last vaccination (Month 6 for the Co-Ad Group, Month 7 for the Control group)
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 523 | 522
Percentage of participants | 4.0 [2.5 to 6.1] | 6.9 [4.9 to 9.4]

14. Secondary Outcome: Percentage of Participants Reporting at Least One Potential Immune-mediated Disease (pIMDs)
Description: pIMDs are a subset of AEs of special interest that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology. The investigator must exercise his/her medical/scientific judgment to determine whether other diseases have an autoimmune origin (i.e., pathophysiology involving systemic or organ-specific pathogenic autoantibodies) and should also be recorded as a pIMD.
Time Frame: From Day 1 until 6 months after last vaccination (Month 6 for the Co-Ad Group, Month 7 for the Control group)
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 523 | 522
Percentage of participants | 0 [0 to 0.7] | 0.6 [0.1 to 1.7]

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected during 7-day follow-up period after each vaccination. Unsolicited AEs were ollected during 30-day follow-up period after each vaccination. SAEs and pIMDs were collected throughout the study period (from Day 1 to study end [6 months after last vaccination]).
Description: Solicited and unsolicited events were reported per participant at any dose for the assessed timeframe (within 30 days after any vaccine dose administration) according to occurence of each event, as pre-specified in Statistical Analysis Plan.
Arm/Group | Co-Ad Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/523 | 6/522
Serious Adverse Events (participants affected / at risk) | 21/523 | 36/522
Other Adverse Events (participants affected / at risk) | 427/523 | 428/522
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-Ad Group (N=523) | Control Group (N=522)
Bronchitis (Infections and infestations) | 2 (3) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Bacterial disease carrier (Infections and infestations) | 1 (1) | 0 (0)
Complicated appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Retroperitoneal abscess (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Superinfection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (5)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Posterior capsule rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound necrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Giant cell arteritis (Vascular disorders) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-Ad Group (N=523) | Control Group (N=522)
Injection site pain (General disorders) | 368 (368) | 349 (496)
Fatigue (General disorders) | 236 (237) | 212 (286)
Injection site erythema (General disorders) | 83 (83) | 76 (84)
Injection site swelling (General disorders) | 67 (67) | 61 (69)
Pyrexia (General disorders) | 14 (14) | 9 (9)
Influenza like illness (General disorders) | 1 (1) | 4 (5)
Administration site erythema (General disorders) | 1 (1) | 0 (0)
Administration site pain (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Vessel puncture site swelling (General disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 201 (203) | 206 (263)
Arthralgia (Musculoskeletal and connective tissue disorders) | 133 (134) | 133 (164)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 167 (167) | 164 (210)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 13 (13) | 15 (17)
COVID-19 (Infections and infestations) | 11 (11) | 14 (14)
Bronchitis (Infections and infestations) | 4 (4) | 5 (5)
Respiratory tract infection (Infections and infestations) | 0 (0) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 4 (4)
Rhinitis (Infections and infestations) | 2 (2) | 3 (3)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Abscess oral (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Immunisation reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Muscle contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 5 (5)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Folate deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Neovascular age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Occult blood positive (Investigations) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT05568797/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/97/NCT05568797/SAP_001.pdf